CLINICAL TRIAL: NCT05902156
Title: The Effect of Electronic Patient Decision Support System Developed for Use Patients with Type 2 Diabetes (DiaPaDeSS) on Self-Management, Patient Activation and Metabolic Parameters
Brief Title: Electronic Patient Decision Support System for Patients with Type 2 Diabetes (DiaPaDeSS)
Acronym: DiaPaDeSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Merve Yuksel, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEK-125
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mobile Health; Type 2 Diabetes; Patient Activation; Self-Management; Decision Support System; Nursing; Randomized Controlled Trial
Keywords: Mobile Health; Type 2 Diabetes; Patient Activation; Decision Support System; Self-Management; Nursing; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Participation

STUDY DESIGN:
Intervention Model Description: Patients with type 2 diabetes will be pretested and randomized (intervention 36, control 36) to the DiaPaDeSS intervention and control groups. Both the DiaPaDeSS intervention and control groups will use the DiaPaDeSS for three months. While participants in the DiaPaDeSS intervention group can reach all contents of the DiaPaDeSS, others can reach only these fields: self-management practice tasks (daily, weekly, quarterly), and measurements questionnaires.
Who Masked: Participant
Masking Description: The participants will be divided into groups according to the randomization list created to assign each patient to a group. Two independent researchers will assign participants to the DiaPaDeSS intervention and control groups and evaluate the outcome measurement data. Researchers will not be blinded because they will perform these interventions. However, the participants will be blinded because they do not know which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DiaPaDeSS intervention group (Experimental): DiaPaDeSS will be introduced to participants with type 2 diabetes during face-to-face interviews. The DiaPaDeSS intervention group will have access to all the contents of the DiaPaDeSS, which includes the patient education information about type 2 diabetes, self-management practice tasks (daily, weekly, quarterly), type 2 diabetes patient education program according to DiaPaDeSS algorithms, and measurement questionnaires. During the follow-up period, the participants in the DiaPaDeSS intervention group will take DiaPaDeSS messages once a week and be reminded to use the education program. The DiaPaDeSS will be asked to use it for three months on daily and weekly inputs. During the follow-up period, the participants can contact the researcher via 24/7 on the DiaPaDeSS. Participants in the DiaPaDeSS intervention group will also receive routine patient education and hospital follow-ups.
  Interventions: Behavioral: DiaPaDeSS
- Control Group (Active Comparator): DiaPaDeSS will be introduced to participants with type 2 diabetes in the control group during face-to-face interviews. The control group will have access to only these fields self-management practice tasks (daily, weekly, quarterly), and measurements questionnaires. The diabetes patient education brochure of the Ministry of Health will be sent to the phones of the active control group in pdf format. Participants in the DiaPaDeSS group will also receive routine patient education and routine hospital follow-up during the three-month follow-up period..
  Interventions: Behavioral: DiaPaDeSS

INTERVENTIONS:
Behavioral: DiaPaDeSS — Web-based mobile health application for patients with type 2 diabetes (the patient education information about type 2 diabetes, self-management practice tasks (daily, weekly, quarterly), type 2 diabetes patient education program according to DiaPaDeSS algorithms, and measurement questionnaires)
  Arms: DiaPaDeSS intervention group
Behavioral: DiaPaDeSS — Web-based mobile health application for patients with type 2 diabetes (only self-management practice tasks (daily, weekly, quarterly), and measurements questionnaires. The diabetes patient education brochure of the Ministry of Health will be sent to the phones of the active control group in pdf format.)
  Arms: Control Group

SUMMARY:
This study evaluates the effects of an electronic patient decision support system developed for the use of patients with type 2 diabetes (DiaPaDeSS) on self-management, patient activation, and metabolic parameters. To manage type 2 diabetes after discharge, patients must continue to perform interventions at home, such as blood glucose monitoring, blood pressure measurement, weight measurement, medication use, and foot care. To achieve this, patient's self-management and activation levels should be increased. This can also lead to positive improvements in the metabolic parameters. It would be beneficial to develop DiaPaDeSS that can increase the self-management and activation levels of patients with type 2 diabetes. The investigators will develop the DiaPaDeSS intervention protocol. Our content includes patient education information about type 2 diabetes, self-management practice tasks (daily, weekly, quarterly), a type 2 diabetes patient education program according to DiaPaDeSS algorithms, and measurement questionnaires. The content of the DiaPaDeSS will be evaluated by 10 experts in the fields of medicine, nursing, and informatics. A feasibility test with seven patients will be conducted to evaluate the usability of DiaPaDeSS. A single-blind, randomized controlled trial design will be used. Patients with type 2 diabetes will be pretested and randomized (intervention 36, control 36) to the DiaPaDeSS intervention and control groups. Both the DiaPaDeSS intervention and control groups will use the DiaPaDeSS for three months. While participants in the DiaPaDeSS intervention group can reach all contents of the DiaPaDeSS, others can reach only these fields: self-management practice tasks (daily, weekly, quarterly), and measurements questionnaires. The effectiveness of the DiaPaDeSS will be evaluated at baseline and at month 3.

DETAILED DESCRIPTION:
Improving patients' self-management is one of the primary goals in the treatment and care of type 2 diabetes. Self-management in patients with type 2 diabetes is recognized as an important factor in controlling blood glucose levels and preventing diabetes-related complications. By strengthening the self-management of patients with type 2 diabetes, positive improvements can be achieved in terms of metabolic parameters. Although the concept of self-management plays an important role in the treatment and care of patients with type 2 diabetes, self-management levels of patients are generally reported to be low. The patients activation levels also affect their ability to maintain self-care and self-management. Patients who are more active tend to participate in self-management behaviors that improve their health. When the relationship between patient activation and self-management was examined, patient activation was associated with better self-management and better health outcomes. Since type 2 diabetes is a common chronic disease, new strategies are needed to improve self-management and activation levels in patients with type 2 diabetes. Decision-support systems are used as a new strategy to provide quality diabetes care. An electronic patient decision support system may help increase patient activation levels, improve self-management levels, and have positive effects on metabolic parameters. It is predicted that the use of electronic patient decision support systems will reduce the frequency of complications, emergency room visits, and health costs in patients with type 2 diabetes. It is thought that an electronic patient decision support system can support the active participation of patients with type 2 diabetes in disease self-management at home. This study evaluates the effect of an electronic patient decision support system developed for self-management, patient activation, and metabolic parameters of patients with type 2 diabetes.

Objective: This study is aimed to develop DiaPaDeSS and evaluate its effects on self-management, patient activation, and metabolic parameters. DiaPaDeSS engages and supports patients with type 2 diabetes by increasing patient activation and self-management through m-health education. This can increase self-management, patient activation, and metabolic parameters. This study primarily aims to analyze the efficacy of DiaPaDeSS in improving self-management, patient activation, and metabolic parameters.

Methods: This study consists of two stages. The first stage of this study was the development of DiaPaDeSS. This stage included reading the content and designing the DiaPaDeSS. The investigators will create the DiaPaDeSS intervention protocol. The DiaPaDeSS content was based on the needs of patients, evidence, and recommendations for patient education in type 2 diabetes, such as guidelines, meta-analyses, randomized controlled trials, reliable national and international patient education websites, and expert opinions. Our content includes patient education information about type 2 diabetes, self-management practice tasks (daily, weekly, quarterly), type 2 diabetes patient education program according to DiaPaDeSS algorithms, and measurement questionnaires. Patient education information topics included diabetes, type of diabetes, signs and symptoms of type 2 diabetes, complications of type 2 diabetes, diagnosis and treatment methods, healthy lifestyle, and enhanced self-management and patient activation. Self-management practice tasks are divided into three groups: daily activity tasks, weekly activity tasks and quarterly activity tasks. Daily activity tasks included blood glucose level monitoring, medication use, and foot care. Weekly activity tasks included taking blood pressure and weight measurements. Quarterly activity tasks included HbA1c, cholesterol, and triglyceride levels at the follow-up. The measurement questionnaires included pre and endpoint questionnaires. The participants can answer the questionnaire via DiaPaDeSS. The content of the DiaPaDeSS will be evaluated by a total of 10 experts in the fields of medicine, nursing and informatics. A feasibility test with seven patients will be conducted to evaluate the usability of the DiaPaDeSS.

In the second stage, the investigators will conduct a single-blind, randomized controlled study to determine the effect of DiaPaDeSS on self-management, patient activation, and metabolic parameters. This study will be conducted in patients with type 2 diabetes who are followed up and treated in the Endocrinology and Metabolic Diseases Polyclinic and who meet the inclusion criteria of the sample. In this study, the sample size was calculated based on Cohen's d effect size coefficient of 0.60, 80% power, and a 5% confidence interval using the G*POWER software package. The study will be conducted in patients with type 2 diabetes (n=72): 36 in the DiaPaDeSS intervention group and 36 in the control group. Patients with type 2 diabetes who had been followed up and treated at the Endocrinology and Metabolic Diseases Polyclinic, aged between 18-65 years, patients who know their diagnosis and can verbally express it, have been diagnosed with type 2 diabetes for at least six months, who are literate, who have internet access at home, who have one of the tools such as a computer, tablet or smartphone and can use these tools, consented to participate in the study, and had no other psychiatric or mental barriers to answering the questions, language or cognitive difficulties, and barriers to verbal or written communication were included. It will be prepared in line with the Consolidated Standards of Reporting Trials (CONSORT 2018) guidelines. There will be screening, pretest at baseline, randomization, and follow-up.

Full sociodemographic and clinical assessments and consent will be obtained during the screening. At the screening stage, all participants will be informed about DiaPaDeSS and this study face to-face at the hospital first. Subsequently, participants could use the DiaPaDeSS at home. The pretest will be carried out at the baseline. Baseline measurements will be undertaken by the researcher before randomization occurs.

As a randomization method, the " stratified block randomization method" will be chosen so that the participants in the intervention (DiaPaDeSS intervention group) and control groups have similar characteristics. During the pretest, patients will be stratified and randomized according to their age, which is considered to be one of the prognostic factors of the study. An independent researcher who was not involved in the research will be assigned to the DiaPaDeSS intervention and control groups using the web-based randomization program. Randomization will be done in http://www.r-bloggers.com/example-2014-2-block-/randomization/ and put in opaque envelopes. The DiaPaDeSS intervention group will have access to all the content of the DiaPaDeSS, which includes the patient education information about type 2 diabetes, self-management practice tasks (daily, weekly, quarterly), type 2 diabetes patient education program according to DiaPaDeSS algorithms, and measurement questionnaires. Passwords will be defined so that patients in the DiaPaDeSS intervention group can access DiaPaDeSS. DiaPaDeSS will be delivered face-to-face at the hospital by the researcher, after which participants could be used at home. Participants in the control group will only have access to the self-management practice tasks (daily, weekly, quarterly), and measurements questionnaires in the DiaPaDeSS. The other fields will be encrypted. Patients in the control group will also be informed of the area that they can access. The DiaPaDeSS intervention group will be asked to use it for three months on daily and weekly input of their self-management practice tasks. The investigators will send a message to participants in the DiaPaDeSS intervention group every week via DiaPaDeSS to remind them of their self-management practice tasks. Participants were blinded because they were unaware of their randomization status. Since the researchers conducted the interventions, it is not possible to blind them to the nature of the study.

The DiaPaDeSS intervention protocol will be prepared specifically for the development of healthy lifestyle behaviors in type 2 diabetes and the prevention or management of acute and chronic complications of type 2 diabetes. The protocol to be developed will be integrated into the website. Within the scope of the intervention protocol, the intervention group will enter the self-management practice task results requested on a daily or weekly basis from the relevant screen to the website. After the requested information is entered, the data will be recorded in the system, and the evaluation will be performed through the algorithms in the knowledge base of the decision support system. As a result of the evaluation, attention and urgent areas will appear on the website screen. According to the results of this evaluation, patient needs will be determined, education on self-management will be displayed through decision-support system algorithms for patient needs, and patients will be guided. Education and guidance will be provided by algorithms designed according to the evaluation results. Patients who do not use DiaPaDeSS will be warned on the website, and in cases where missing registration data are detected despite the warning, reminders will be made by calling them via SMS and/or phone. Participants in the control group will only have access to the self-management practice tasks (daily, weekly, quarterly), and measurements questionnaires in the DiaPaDeSS. The diabetes patient education brochure of the Ministry of Health will be sent to the phones of the active control group in pdf format. They will also receive routine patient education and hospital follow-ups.

Primary outcomes are self-management, patient activation, and metabolic parameters. Outcomes will be measured at baseline and follow-up, occurring 3 months after enrolment. The hypotheses are as follows:

It is hypothesized that, compared with those receiving standard care after controlling for baseline levels, participants receiving the DiaPaDeSS intervention will report significantly.

1. Participants receiving the DiaPaDeSS intervention will have higher levels of self-management than those receiving standard care, after controlling for baseline levels of self-management.
2. Participants receiving the DiaPaDeSS intervention will have higher levels of patient activation than those receiving standard care, after controlling for baseline levels of patient activation.
3. Participants receiving the DiaPaDeSS intervention will have improved metabolic parameters (a) HbA1c, b) blood glucose, c) blood pressure, d) cholesterol, e) triglyceride levels, and f) body mass index) than those receiving standard care after controlling for baseline levels of metabolic parameters.

The investigators will evaluate the outcomes using the Type 2 Diabetes Self-Management Scale, Patient Activation Measure (PAM), and Metabolic Parameter Monitoring Form.

Primary Outcome Measures Type 2 Diabetes Self-Management Scale: The Type 2 Diabetes Self-Management Scale was developed to evaluate the self-management of patients with type 2 diabetes. The scale consists of 19 items and three sub-dimensions. These dimensions were determined as the "Healthy Lifestyle Behaviors" dimension consisting of 11 questions, the "Health Services Use" dimension consisting of four questions, and the "Blood Sugar Management" dimension consisting of four questions. Scoring of the scale: "always 5 points", "often 4 points", "sometimes 3 points", "rarely 2 points", and "never 1 point". High scores on the scale indicate good self-management, whereas low scores indicate poor self-management. Cronbach's alpha for the scale was determined as 0.85.

Patient Activation Measure (PAM): The Patient Activation Measure (PAM) gauges a patient's level of belief, knowledge, skill, and self-assurance. Thirteen components comprise the Patient Activation Measure. Patients actively and successfully managed their disease when they received higher scores on the scale. Each response option has a 4-point Likert scale with the options ranging from totally disagree to totally agree and non applicable. The scores for the activities ranged from 0 to 100. Level 1, the lowest activity with a score of 47, deals with the idea that playing an active role is important. Level 2, which ranges from 47 to 55, denotes the knowledge and capacity for action. Level 3, which ranges from 55 to 72, deals with actions. The highest activity, Level 4, with scores >72.5, was maintained at a Schedule even under stress. Cronbach's alpha value of the original scale was 0.88.

Metabolic Parameter Monitoring Form: The Metabolic Parameter Monitoring Form was created by researchers in line with the literature to evaluate the results that may affect the prognosis of type 2 diabetes during the application process. It was created to evaluate the changes in basic parameters (HbA1c, blood glucose, blood pressure, cholesterol, triglyceride values, body mass index) that should be evaluated in patients with type 2 diabetes. In the first meeting, we planned to obtain the laboratory results of the patients from the electronic patient records with the permission of the diabetes nurses in the Endocrinology and Metabolic Diseases Polyclinic, and to compare them with the laboratory results last examined at the end of the third month.

Conclusion: DiaPaDeSS is expected to improve self-management, patient activation, and metabolic parameters in patients with type 2 diabetes. This study could contribute to the innovation of healthcare by developing a new digital tool for patient education.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes who had been followed up and treated at the Endocrinology and Metabolic Diseases Polyclinic
* Aged between 18-65 years
* Patients who know their diagnosis and can verbally express it
* Have been diagnosed with type 2 diabetes for at least six months
* Who are literate
* Who have internet access at home, who have one of the tools such as a computer, tablet or smartphone and can use these tools
* Consented to participate in the study
* Had no other psychiatric or mental barriers to answering the questions, language or cognitive difficulties, and barriers to verbal or written communication

Exclusion Criteria:

* Diagnosed with myocardial infarction, stroke or diabetic foot in the last six months
* Diagnosed with type 1 diabetes or gestational diabetes
* Diagnosed with terminal illness
* Using steroid therapy
* Had pregnant
* Having dementia and cognitive deficits
* Having retinopathy or advanced neuropathy
* Patients whose information is not allowed to be accessed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The Type 2 Diabetes Self-Management Scale | 12 weeks
  The Type 2 Diabetes Self-Management Scale was developed to evaluate the self-management of patients with type 2 diabetes. The scale consists of a total of 19 items and three sub-dimensions. These dimensions were determined as the "Healthy Lifestyle Behaviors" dimension consisting of 11 questions, the "Health Services Use" dimension consisting of four questions, and the "Blood Sugar Management" dimension consisting of four questions. Scoring of the scale; "always 5 points", "often 4 points", "sometimes 3 points", "rarely 2 points", "never 1 point". High scores on the scale indicate good self-management, and low scores indicate poor self-management. The Cronbach's alpha value of the scale was determined as 0.85.
Patient Activation Measure (PAM) | 12 weeks
  The Patient Activation Measure (PAM) gauges a patient's level of belief, knowledge, skills, and self-assurance. Thirteen components comprise the Patient Activation Measure. Patients are actively/successfully managing their disease when they receive higher scores on the scale. Each response option has a 4-point Likert scale with the options ranging from totally disagree to totally agree and 'non applicable.' Scores for activities range from 0 to 100. Level 1, the lowest activity with a score of 47, deals with the idea that playing an active part is important. Level 2, which ranges from 47 to 55, denotes knowledge and the capacity for action. Level 3, which ranges from 55 to 72, deals with action. The highest activity, Level 4, with scores of >72.5, is keeping to a Schedule even when under stress. Cronbach's alpha value of the original scale was determined as 0.88.
The Metabolic Parameter Monitoring Form | 12 weeks
  The Metabolic Parameter Monitoring Form was created by researchers in line with the literature to evaluate results that may affect the prognosis of type 2 diabetes during the application process. It was created to evaluate the changes in the basic parameters: (a) HbA1c (mmol/L), (b) blood glucose (mg/dL), (c) blood pressure (mmHg), (d) cholesterol (mg/dL), (e) triglyceride (mg/dL) values, (f) body mass index ((weight and height will be combined to report BMI in kg/m2) that should be evaluated in patients with type 2 diabetes. In the first meeting, it is planned to obtain the laboratory results of the patients from the electronic patient records with the permission of the diabetes nurses in the Endocrinology and Metabolic Diseases Polyclinic and to compare them with the laboratory results last examined at the end of the third month. Average value will be calculated for levels taken in the first and last month.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
This can be shared privately if other researchers wish to obtain it.